CLINICAL TRIAL: NCT07386262
Title: Efficacy and Safety of the Adacolumn® Granulocyte and Monocyte/Macrophage Apheresis Device for Cerebral Edema After Acute Anterior Circulation Occlusive Cerebral Infarction: A Prospective, Randomized, Controlled Clinical Trial
Brief Title: A Trial of Adacolumn on Cerebral Edema After Anterior Circulation Ischemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-1867
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Edema; Ischemic Stroke, Acute; Malignant Cerebral Edema; Anterior Circulation Brain Infarction
MeSH Terms: conditions — Brain Edema; Ischemic Stroke; Brain Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Device: Adacolumn® (Experimental): Adacolumn Treatment Combined with Endovascular Thrombectomy and Standard Medical Therapy
  Interventions: Device: Adacolumn®; Procedure: Endovascular Thrombectomy; Drug: Standard medical management
- Standard Treatment (Active Comparator): Endovascular Thrombectomy and Standard Medical Therapy
  Interventions: Procedure: Endovascular Thrombectomy; Drug: Standard medical management

INTERVENTIONS:
Device: Adacolumn® — Adacolumn treatment ：once a day for 4 consecutive days after enrollment (60 minutes each time, blood flow rate 30 mL/min, total blood volume processed 1800 mL); the treatment was performed by establishing extracorporeal circulation through bilateral arm veins, and a total of 4 adsorption treatments were completed.
  Arms: Device: Adacolumn®
Procedure: Endovascular Thrombectomy — Endovascular thrombectomy will be performed in strict accordance with the indications, contraindications, and operational specifications outlined in the Chinese Stroke Society Guidelines for Reperfusion Therapy in Acute Ischemic Stroke (2024), as well as the latest official instructions for use of the relevant endovascular devices and adjunctive medications.
Drug: Standard medical management — Standard medical management for ischemic stroke.

SUMMARY:
The primary objective is to investigate whether treatment with Adacolumn can ameliorate the progression of cerebral edema within 72 hours in patients with anterior circulation ischemic stroke. The secondary objective is to explore if Adacolumn could improve acute neurologic status, functional outcomes, treatment requirements and safety in patients with anterior circulation ischemic stroke.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled trial evaluating Adacolumn therapy in patients with acute ischemic stroke due to anterior circulation large-artery occlusion presenting within 10 hours of stroke onset. Eligible patients who meet all inclusion and no exclusion criteria will be randomized in a 1:1 ratio to the Adacolumn group or the control group, with 5 patients enrolled in each arm (total n=10).

All participants will have undergone guideline-based endovascular thrombectomy for acute ischemic stroke, together with standard medical management. In the Adacolumn group, each patient will undergo four scheduled Adacolumn treatment sessions in addition to endovascular thrombectomy and standard medical therapy. Patients in the control group will receive endovascular thrombectomy and standard medical treatment alone. Each participant will be followed for 90 days after enrollment.

The objective of the trial is to evaluate the effect of Adacolumn therapy on cerebral edema in patients with anterior circulation large-artery occlusion stroke. The primary endpoint is the change in net water uptake (NWU) measured on CT at 72-78 hours post reperfusion, compared to the immediate post-reperfusion CT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, regardless of gender;
2. A clinical diagnosis of acute ischemic stroke;
3. Proven large vessel occlusion in ICA or MCA-M1 occlusion (carotid occlusions can be cervical or intracranial, with or without tandem MCA lesions) determined by MRA or CTA or DSA;
4. NIHSS score ≥10 at screening;
5. Pre-stroke mRS score <2 (independent in all activities of daily living);
6. Time from stroke onset to initiation of the first Adacolumn treatment is ≤10 hours, stroke onset is defined as the last time the patient was known to be at their neurological baseline (wake-up strokes qualify if within this time window);
7. All endovascular thrombectomy procedures must strictly adhere to the "2024 Chinese Stroke Association Guidelines for Reperfusion Therapy in Acute Ischemic Stroke" and the latest prescribing information/instructions for use regarding indications, contraindications, and procedural standards;
8. Written informed consent obtained from the patient or legally authorized representative.

Exclusion Criteria:

1. Decompressive craniectomy performed before enrollment or between enrollment and initiation of study treatment;
2. Patients who receive intravenous thrombolysis (including bridging therapy) for the index ischemic stroke episode before or during endovascular thrombectomy; or undergo permanent intracranial or extracranial stent implantation (including intracranial stent-assisted thrombectomy or carotid stenting) during the index endovascular procedure;
3. After endovascular thrombectomy: extensive contrast extravasation (diffuse subarachnoid high density or parenchymal high density not consistent with hematoma), new subarachnoid hemorrhage（SAH）, or symptomatic intracranial hemorrhage (sICH);
4. Large-vessel occlusion is attributed to other determined etiologies per TOAST classification, such as tumor-related, dissection-related, or other clearly identifiable non-LAA/non-CE causes.
5. Clinical signs of brain herniation, such as unilateral or bilateral fixed dilated pupils and/or other loss of brainstem reflexes attributable to cerebral edema or herniation in the investigator's opinion;
6. Intracranial lesions conferring markedly increased bleeding risk (known brain tumor, arteriovenous malformation, aneurysm);
7. Inability to undergo MRI;
8. Absolute neutrophil count <1.5×10⁹/L or >15×10⁹/L
9. Absolute monocyte count > 1.0 ×10⁹/L;
10. Red blood cells <3.0×10¹²/L ;
11. Active internal bleeding or bleeding tendency (such as platelet count <100×10⁹/L, INR >1.7, PT >15 seconds);
12. Marked hypercoagulability (fibrinogen >700 mg/dL);
13. Intracranial or spinal surgery or severe head trauma within the past 3 months;
14. Refractory hypertension (persistent systolic blood pressure >185 mmHg or diastolic >110 mmHg);
15. Known allergy to components of the blood purification system (including adsorption membrane, anticoagulants);
16. Acute ST-segment elevation myocardial infarction and/or acute decompensated heart failure and/or corrected QT interval >520 ms and/or history of cardiac arrest within the past 6 months(pulseless electrical activity, ventricular tachycardia, ventricular fibrillation, or asystole);
17. Body temperature >38°C or active infection;
18. Active autoimmune disease or immunodeficiency;
19. Participation in another interventional clinical trial within the past 30 days;
20. Any other condition deemed unsuitable for participation by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in net water uptake (NWU) on CT between the immediate post-reperfusion and 72-78 hours post-reperfusion | 72 hours
  The change in net water uptake (NWU) measured on CT at 72-78 hours post-reperfusion, compared to the immediate post-reperfusion CT

SECONDARY OUTCOMES:
Serious adverse events (SAEs) related to Adacolumn treatment (Primary Safety Outcome) | Randomization to Day 90
  Adacolumn treatment-related SAEs specifically including but not limited to: hypotension requiring vasopressor support (systolic blood pressure <90 mmHg); access site hemorrhage or hematoma; infection (manifested as fever or access site erythema); electrolyte disturbances such as hypokalemia or hypocalcemia; thrombocytopenia (platelet count <100 × 10⁹/L); and any other event judged by the investigator to be a treatment-related SAE.
The number of discontinuation of Adacolumn therapy due to adverse events (Safety Outcome) | Randomization up to Day 3
  Record the number of patients who permanently discontinued Adacolumn therapy during the treatment period specifically due to SAEs
The change in midline shift on CT between the immediate post-reperfusion and 72-78 hours post-reperfusion | 72 hours
Change in National Institutes of Health Stroke Scale (NIHSS) score on day 7 post-treatment compared to immediate post-operative baseline | Day 7
Number of participants who developed brain herniation after treatment | Baseline up to Day 14
Number of participants who underwent decompressive craniectomy (DC) | Baseline up to Day 14
modified Rankin Scale (mRS) Score | Day 90
Number of participants who achieved mRS 0-2 | Day 90
Number of participants who achieved mRS 0-3 | Day 90
Number of participants with death | Baseline up to Day 90
The relative percentage change in DWI edema volume at day 4 post-reperfusion compared to the immediate post-reperfusion DWI | Day 4
The relative percentage change in DWI infarct volume at day 4 post-reperfusion compared to the immediate post-reperfusion DWI | Day 4

OTHER OUTCOMES:
Dynamic changes in peripheral blood immune cells before and after Adacolumn therapy | Baseline up to Day 3、 Day 7
Cerebral immune cell infiltration analysis | Baseline up to Day 14
  For patients undergoing decompressive craniectomy combined with internal decompression, intraoperative brain tissue samples will be collected from the infarct region. These specimens will be subjected to comprehensive analysis to characterize the infiltration, including quantification, phenotypic identification, and functional assessment of immune cells

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dignass A, Akbar A, Hart A, Subramanian S, Bommelaer G, Baumgart DC, Grimaud JC, Cadiot G, Makins R, Hoque S, Bouguen G, Bonaz B. Safety and Efficacy of Granulocyte/Monocyte Apheresis in Steroid-Dependent Active Ulcerative Colitis with Insufficient Response or Intolerance to Immunosuppressants and/or Biologics [the ART Trial]: 12-week Interim Results. J Crohns Colitis. 2016 Jul;10(7):812-20. doi: 10.1093/ecco-jcc/jjw032. Epub 2016 Jan 27. PMID 26818659
- [Background] Elkins J, Veltkamp R, Montaner J, Johnston SC, Singhal AB, Becker K, Lansberg MG, Tang W, Chang I, Muralidharan K, Gheuens S, Mehta L, Elkind MSV. Safety and efficacy of natalizumab in patients with acute ischaemic stroke (ACTION): a randomised, placebo-controlled, double-blind phase 2 trial. Lancet Neurol. 2017 Mar;16(3):217-226. doi: 10.1016/S1474-4422(16)30357-X. Epub 2017 Feb 15. PMID 28229893
- [Background] Ren T, Zhu M, Jiang X, Xu L, Jin H, Zhou Y, Zhao Y, Zhuo R, Li W, Chen C, Peng L, Jin X, Li Y, Yang L. Targeting microglial PPARalpha ameliorates the outcome of ischemic stroke by enhancing interaction with infiltrating peripheral monocytes/macrophages. Cell Rep. 2025 Jul 22;44(7):115875. doi: 10.1016/j.celrep.2025.115875. Epub 2025 Jun 20. PMID 40543039
- [Background] Shi K, Tian DC, Li ZG, Ducruet AF, Lawton MT, Shi FD. Global brain inflammation in stroke. Lancet Neurol. 2019 Nov;18(11):1058-1066. doi: 10.1016/S1474-4422(19)30078-X. Epub 2019 Jul 8. PMID 31296369
- [Background] Huttner HB, Schwab S. Malignant middle cerebral artery infarction: clinical characteristics, treatment strategies, and future perspectives. Lancet Neurol. 2009 Oct;8(10):949-58. doi: 10.1016/S1474-4422(09)70224-8. PMID 19747656
- [Background] Wu S, Yuan R, Wang Y, Wei C, Zhang S, Yang X, Wu B, Liu M. Early Prediction of Malignant Brain Edema After Ischemic Stroke. Stroke. 2018 Dec;49(12):2918-2927. doi: 10.1161/STROKEAHA.118.022001. PMID 30571414
- [Background] Sheth KN, Petersen NH, Cheung K, Elm JJ, Hinson HE, Molyneaux BJ, Beslow LA, Sze GK, Simard JM, Kimberly WT. Long-Term Outcomes in Patients Aged </=70 Years With Intravenous Glyburide From the Phase II GAMES-RP Study of Large Hemispheric Infarction: An Exploratory Analysis. Stroke. 2018 Jun;49(6):1457-1463. doi: 10.1161/STROKEAHA.117.020365. Epub 2018 May 22. PMID 29789393
- [Background] Huang X, Yang Q, Shi X, Xu X, Ge L, Ding X, Zhou Z. Predictors of malignant brain edema after mechanical thrombectomy for acute ischemic stroke. J Neurointerv Surg. 2019 Oct;11(10):994-998. doi: 10.1136/neurintsurg-2018-014650. Epub 2019 Feb 23. PMID 30798266